CLINICAL TRIAL: NCT02118181
Title: Role of Oral Supplementation of Proteins and β-hydroxy-β-methyl Butyrate (HMB) in a Sample of Older Women in Good Health
Brief Title: Assessment of Physical Performance With A Supplementation Containing HMB in a Sample of Old Women in Good Health
Acronym: HMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Giuseppe Sergi, Dr, PhD, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Not Avalaible
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-04

CONDITIONS: Age Related Muscle Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- HMB (Experimental): Group taking oral supplementation with Beta-hydroxy-beta-methylbutyrate
  Interventions: Dietary Supplement: HMB

INTERVENTIONS:
Dietary Supplement: HMB
  Arms: HMB

SUMMARY:
The purpose of this study is to determine whether a supplementation containing β-Hydroxy-β-methylbutyrate is effective in the treatment of age-related muscle loss in a group of older women compared to a non interventional group

ELIGIBILITY:
Inclusion Criteria:

* People over 65 years, not residents in nursing home, in good health
* Mini Mental State Examination (corrected for scholarity) more than 23

Exclusion Criteria:

* Previous oral supplementation with proteins or minerals
* important co-mordidities, such renal or hepatic failure

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery | Baseline and after 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Sergi, MD, Principal Investigator — University of Padova
Locations (1):
- University of Padova, Padua, Padua, Italy

REFERENCES:
- [Derived] Berton L, Bano G, Carraro S, Veronese N, Pizzato S, Bolzetta F, De Rui M, Valmorbida E, De Ronch I, Perissinotto E, Coin A, Manzato E, Sergi G. Effect of Oral Beta-Hydroxy-Beta-Methylbutyrate (HMB) Supplementation on Physical Performance in Healthy Old Women Over 65 Years: An Open Label Randomized Controlled Trial. PLoS One. 2015 Nov 3;10(11):e0141757. doi: 10.1371/journal.pone.0141757. eCollection 2015. PMID 26529601